CLINICAL TRIAL: NCT00274092
Title: A Comparison of 18 Mcg of Tiotropium Inhalation Capsules and Atrovent Metered Dose Inhaler (2 Puffs of 20 Mcg) in a Double-Blind, Double-Dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Tiotropium Inhalation Capsules and Atrovent MDI in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.279
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: tiotropium inhalation capsules (18 mcg once daily)
Drug: Atrovent MDI (2 puffs of 20 mcg(q.i.d.) in patients

SUMMARY:
The objective of this study is to compare the bronchodilator efficacy and safety of tiotropium inhalation capsules (18 mcg once daily) and Atrovent MDI (2 puffs of 20 mcg q.i.d.) in patients with chronic obstructive pulmonary disease (COPD)

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, parallel group study to compare the bronchodilator efficacy and safety of tiotropium inhalation capsules and Atrovent MDI in patients with chronic obstructive pulmonary disease (COPD).

Following an initial screening visit, patients will enter a 2-week baseline period. Patients who successfully complete this phase will be randomized into the double-blind portion of the study in which they will receive tiotropium once daily (morning) or Atrovent four times daily. Pulmonary function testing will be conducted just prior to the start of therapy at Visit 2 (i.e. randomization visit after completion of the 2-week run-in period) and at 120 minutes post-dosing. Pulmonary function testing will be repeated at the same time intervals at the end of therapy.

Study Hypothesis:

Null and alternative hypotheses The primary objective of this study was addressed by a two-sided test at the 0.05 level of significance of the null hypothesis that, in patients with chronic obstructive pulmonary disease (COPD), the bronchodilator efficacy after one month is no greater on tiotropium inhalation capsules (18mcg once daily) than on ATROVENT MDI (2 puffs of 20 mcg q.i.d.), against the alternative hypothesis that the bronchodilator efficacy is greater on tiotropium inhalation capsules (18 mcg once daily).

Comparison(s):

Trough FEV1 response will be analyzed. Peak FEV1, FVC trough and peak response, number of Rescue Medication and change from baseline in total score of Patient Evaluation Questionnaire will be analyzed. Change from baseline in each category score of Patient Evaluation Questionnaire will be also analyzed.

ELIGIBILITY:
Inclusion:

1. COPD patients with an Forced Expiratory Volume in one second (FEV1)<= 65% of predicted normal and FEV1 <= 70% of Forced Vital Capacity (FVC).
2. Male or female patients 40 years of age or older.
3. Patients must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year.
4. Patients must be able to perform pulmonary function tests as required in the protocol.
5. Patients must be able to inhale medication from the HandiHaler device and should have a good technique of inhaling aerosol administered from an MDI..
6. All patients must sign an Informed Consent Form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications.

Exclusion:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded.
3. All patients with a SGOT and SGPT twice the upper normal limit, bilirubin 150% or creatinine 125% of the upper normal limit will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these subjects.
4. Patients with a recent history (i.e. one year or less) of myocardial infarction.
5. Any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
6. Patients with regular use of daytime oxygen therapy.
7. Patients with known active tuberculosis.
8. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed.
9. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
10. A history of thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per Exclusion 1.
11. Patients with an upper respiratory tract infection in the past 6 weeks prior to the Screening Visit (=Visit 1) or during the baseline period of 2-weeks (run-in period).
12. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other component of the inhalation capsule delivery system.
13. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction. (Patients on BPH medications with minimum symptoms are permitted).
14. Patients with known narrow-angle glaucoma.
15. Patients who are being treated with cromolyn sodium or nedocromil sodium.
16. Patients who are being treated with antihistamines.
17. Patients using oral corticosteroid medication at unstable dosage (i.e. less than 6 weeks on a stable dose) or at a dose in excess of the equivalent 10 mg of prednisone per day or 20 mg every other day.
18. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices, or diaphragm).
19. Patients with a history of asthma, allergic rhinitis or atopy or who have a blood total eosinophil count bigger or equal 400 per ul (males) or bigger/equal 320 per ul (females). A repeat eosinophil count will not be conducted in these patients.
20. Patients with a history and/or active alcohol or drug abuse.
21. Patients who have taken an investigational drug one month or six half-lives (whichever is greater) prior to the Screening Visit (=Visit 1).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2002-09; Primary Completion 2003-10 (Actual); Study Completion 2003-10

PRIMARY OUTCOMES:
The primary endpoint is trough FEV1 response which is defined as change from baseline FEV1 (visit 2) and trough FEV1 at week 4 (visit 4)

SECONDARY OUTCOMES:
FEV1 and FVC response at 2 hours post drug administration at on each pulmonary test day; Trough FVC response; Number of rescue medications; and Change from baseline in total score of patient evaluation questionnaire at week 4 (visit 4).

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Taiwan Ltd.
Locations (6):
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Veterans General Hospital, Taipei